CLINICAL TRIAL: NCT06525012
Title: Observational Study on Mortality and Outcome of Patients Hospitalized for Subarachnoid Hemorrhage of Aneurysmal Origin in Martinique Between 2013 and 2021
Acronym: HSA Rankin
Status: Recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 24_RIPH3-01
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Subarachnoid Hemorrhage of Aneurysmal Cause
Keywords: SAH (Subarachnoid Hemorrhage); Ruptured intracranial aneurysm; Modified Rankin score; Mortality; Patient autonomy; Patient dependence
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SAH of aneurysmal origin in hospitalized patients in Martinique between 2013 and 2021
  Interventions: Other: Usual patient care for patients hospitalized for subarachnoid hemorrhage of aneurysmal origin

INTERVENTIONS:
Other: Usual patient care for patients hospitalized for subarachnoid hemorrhage of aneurysmal origin — During hospitalization (2013-2021), patients were managed after multidisciplinary consultation in accordance with national recommendations between resuscitators, neurosurgeons and neuroradiologists, depending on the severity of the initial management and the patient's comorbidities, either by interventional radiology, neurosurgery or medical treatment.

SUMMARY:
The aim of our study is to analyze mortality and sequelae of subarachnoid hemorrhage of aneurysmal origin in hospitalized patients in Martinique. Predictive factors of poor prognosis will also be analyzed.

DETAILED DESCRIPTION:
Subarachnoid hemorrhage is an uncommon pathology in the general population, with a worldwide incidence of 9 per 100,000 people/year, but with a non-negligible risk of sequelae in terms of impairments, activity limitations and participation restrictions of around 30%. Mortality remains high at 40%, despite increasingly specialized care.

In addition, there are a number of objective, rapid assessment scores for autonomy and impairments, notably the modified Rankin score, which is not specific to subarachnoid hemorrhage, but which enables the study of patients' perceived quality of life. Certain factors predictive of bad patient outcome are known in the literature, but have been little studied in the population of Martinique.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) patients,
* Admitted to University Hospital of Martinique with subarachnoid hemorrhage of aneurysmal origin between 01/01/2013 and 31/12/2021,
* Informed patient/next-of-kin/treating physician consent for research participation.

Exclusion Criteria:

* Other causes of subarachnoid hemorrhage of non-aneurysmal origin (traumatic, arteriovenous malformation, cerebral tumor, cerebral thrombophlebitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Martinique for subarachnoid hemorrhage of aneurysmal origin
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate mortality in patients hospitalized for subarachnoid hemorrhage of aneurysmal origin over a 9-year period (2013-2021) in Martinique. | 6 months
  Mortality of subarachnoid hemorrhage of aneurysmal origin.

SECONDARY OUTCOMES:
Evaluate the clinical outcome of these patients. | 6 months
  Patient's clinical outcome (mortality, impairment of patient autonomy, impairment of patient's level of dependece), assessed with the modified Rankin score at discharge and at a distance from hospitalization (minimum delay: 2.5 years).
Analyze the factors associated with a significant impairment of autonomy and/or dependence. | 6 months
  Predictive factors associated with significant impairment of patient autonomy and/or dependence (modified Rankin score = 4 or 5): age, degree of consciousness at the time of treatment (WFNS score), amount of blood in the meningeal spaces (Fisher score), aneurysm size
Analyze the factors associated with death. | 6 months
  Predictive factors associated with death (modified Rankin score = 6): age, degree of consciousness at the time of treatment (WFNS score), amount of blood in the meningeal spaces (Fisher score), aneurysm size.
Analyze the factors associated with a poor prognosis (death AND/OR significant impairment of autonomy/dependence). | 6 months
  Predictive factors associated with a poor prognosis (modified Rankin score ≥ 4: death AND/OR impaired patient autonomy and/or dependence): age, degree of consciousness at the time of treatment (WFNS score), amount of blood in the meningeal spaces (Fisher score), aneurysm size.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No